CLINICAL TRIAL: NCT04504136
Title: Regulation of Mucosal Healing in Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terrence A Barrett (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Terrence A Barrett, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IMDDN-20-MUCOSALHEALING; 2R01DK095662-10A1 (NIH)
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: mucosal; rheumatoid arthritis; psoriatic arthritis; ulcer; colitis; Crohn's; mitochondria; biopsy; wound; biologic; anti-TNF
MeSH Terms: conditions — Inflammatory Bowel Diseases; Arthritis, Rheumatoid; Arthritis, Psoriatic; Ulcer; Colitis; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Controls (Experimental): Participants in this group will be healthy (not diagnosed with inflammatory bowel disease).
  Interventions: Procedure: Serial Biopsy
- Inflammatory Bowel Disease (Experimental): Participants in this group will have been diagnosed with ulcerative colitis (UC) or Crohn's disease (CD) and have either failed treatment with biologics or be naive to biologic therapy.
  Interventions: Procedure: Serial Biopsy
- Rheumatoid/Psoriatic Arthritis (Experimental): Participants in this group will have been diagnosed with rheumatoid (RA) or psoriatic arthritis (PsA) and will be receiving anti-TNF antibody therapy at the time of enrollment.
  Interventions: Procedure: Serial Biopsy

INTERVENTIONS:
Procedure: Serial Biopsy — During the initial colonoscopy, 16-20 biopsies will be collected in addition to standard of care biopsies, and biopsy sites will be tattoed. Patients will return for a follow-up colonoscopy 4-35 days later. An additional 16-20 biopsies will be collected in a "biopsy of the biopsy" approach.

SUMMARY:
The objective of the current study is to compare non-healing colonic ulcers in patients with inflammatory bowel disease (IBD) with iatrogenic colonic ulcers (biopsy sites) in healthy control patients and patients with rheumatoid or psoriatic arthritis. Patients will be biopsied at baseline and again at a follow-up visit in a "biopsy of the biopsy" approach. These biopsies will be used to reveal patterns about gene expression and mitochondrial function during ulcer healing.

DETAILED DESCRIPTION:
Induction of mucosal healing in inflammatory bowel disease (IBD) is associated with reduced hospitalizations, surgeries, and reduced cancer risk. However, previous studies have shown that 54-69% of ulcerative colitis (UC) patients fail to heal ulcers after several weeks of treatment, and roughly half do not maintain remission at one year. The single most important factor in preventing severe medical consequences, like colon removal surgery or cancer, is treatment to completely heal the top layer of the intestine as quickly as possible. Healing is a complex process and the dysfunction observed in colitis can only be fully understood by comparison to healing in non-IBD patients.

This is a prospective trial involving three groups of patients: 1) IBD patients with active disease, newly treated with anti-TNF therapy (biologic failure or naïve); 2) non-IBD patients with rheumatoid/psoriatic arthritis who are receiving anti-TNF therapy, and 3) healthy control patients. Biopsies will be collected at baseline during standard of care endoscopy and at a follow-up research endoscopy.

This study will probe mechanisms of ulcer healing by analyzing gene expression patterns and mitochondrial function.

ELIGIBILITY:
Inclusion Criteria (Group 1):

* Diagnosed ulcerative colitis or Crohn's disease
* Biologic failure or naive to biologic treatment
* Eligible to be treated with anti-TNF therapy

Inclusion Criteria (Group 2):

* Diagnosed rheumatoid or psoriatic arthritis
* Receiving anti-TNF antibody therapy at the time of enrollment

Inclusion Criteria (Group 3):

* Endoscopically unremarkable colonic mucosa
* Absence of inflammatory bowel disease

Exclusion Criteria:

* Classified in an anesthesia risk group, ASA Class =4
* History of bleeding diathesis or coagulopathy
* Stroke or transient neurological attack with the last 6 months
* Pregnant
* Receiving anticoagulants or anti-platelet medications other than low-dose aspirin
* Receiving steroid therapy or metformin
* HIV positive
* Incarceration
* History of total proctocolectomy
* History of system chemotherapy within 18 months
* Uncontrolled intercurrent illness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial DNA copy number | 35 days
  Mitochondrial DNA copy number will be measured in epithelial cells collected from biopsies taken during the initial colonoscopy and at the follow-up colonoscopy.
Change in expression levels of cMyc | 35 days
  Relative expression of cMyc (mRNA) will be measured in epithelial cells collected from biopsies taken during the initial colonoscopy and at the follow-up colonoscopy.
Change in expression levels of PGC-1 alpha | 35 days
  Relative expression of PGC-1 alpha (mRNA) will be measured in epithelial cells collected from biopsies taken during the initial colonoscopy and at the follow-up colonoscopy.
Change in expression levels of Ki67 | 35 days
  Relative expression of Ki67 alpha (mRNA) will be measured in epithelial cells collected from biopsies taken during the initial colonoscopy and at the follow-up colonoscopy.
Number of visible ulcers | 1 day (at follow-up visit)
  The number of visible ulcers will be assessed during the follow-up endoscopy for healthy patients and rheumatoid/psoriatic arthritis patients only.

SECONDARY OUTCOMES:
Change in Mayo Endoscopic Score | 35 days
  The Mayo Endoscopic Score will be calculated at baseline and at follow-up in patients with ulcerative colitis only. The Mayo Endoscopic score is evaluated for the macroscopically most severely inflamed segment: 0 for normal or inactive disease; 1 for erythema, decreased vascular pattern, mild friability; 2 for marked erythema, absent vascular pattern, friability, erosions; 3 ulcerations or spontaneous bleeding. Segmental scores range from 0-3; higher scores indicate more severe disease.
Change in Segmental SES-CD Score | 35 days
  The Simple Endoscopic Score (SES) will be calculated at baseline and follow-up in patients with Crohn's disease (CD) only. The SES-CD score incorporates ulcer size, narrowing, and the area affected by disease or ulceration. Scores range from 0-12; lower scores indicate remission while higher scores indicate severe endoscopic activity.

OTHER OUTCOMES:
Fecal calprotectin levels | 35 days
  Levels of fecal calprotectin (ug/g) will be measured from stool samples collected from patients at any time during the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Barrett, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No